CLINICAL TRIAL: NCT05206331
Title: Contrast Enhanced Mammography (CEM) to Reduce Biopsy Rates for Less Than Highly Suspicious Breast Abnormalities: a Prospective Study
Brief Title: CEM to Reduce Biopsy Rates for Less Than Highly Suspicious Breast Abnormalities: a Prospective Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Margarita Louise Zuley (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Margarita Louise Zuley, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY21070030; 1R01CA258898 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-25 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: eligible participants will have contrast enhanced mammography before their scheduled biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- contrast enhanced mammography (Experimental): Women who have been recently diagnosed with a suspicious abnormality for which they have scheduled a breast biopsy and meet inclusion criteria will be invited to have a contrast enhanced mammography before their scheduled biopsy procedure.
  Interventions: Device: contrast enhanced mammography; Drug: Iodinated Contrast Media (ICM)

INTERVENTIONS:
Device: contrast enhanced mammography — Dual-energy contrast images; low-energy CEM images will be obtained with a kilovoltage below 35 kVp while the high-energy images will be obtained with 45-49 kVp.The average glandular dose of the CEM procedure is approximately 2.44 mGy per view
Drug: Iodinated Contrast Media (ICM) — standard FDA-approved low osmolarity Iodine contrast agent with 350-370 mg/ml

SUMMARY:
One of the primary criticisms of mammography is that it leads to unneeded stress and anxiety from identification and biopsy of non-cancerous findings. Contrast-enhanced mammography (CEM) has the potential to significantly reduce biopsy rates for commonly seen benign breast lesions while preserving very high cancer detection. The investigators propose a prospective clinical study of patients with diagnostic mammograms rated as BIRADS 4A or 4B and scheduled for a biopsy, in which, prior to undergoing their scheduled biopsy, a CEM procedure is performed. The investigators will test the primary hypothesis that for soft tissue lesions (i.e. masses, asymmetries, architectural distortions) initially rated BI-RADS 4A/4B adding CEM will reduce, by at least 20%, the number of biopsy recommendations for actually benign cases and, at the same time, provide a negative predictive value (NPV) higher than 95%.

DETAILED DESCRIPTION:
The investigators believe that an operationally simple, cost effective, contrast enhanced mammogram (CEM), performed during the patient's diagnostic evaluation, would be the best approach to improve the accuracy of radiologists' decisions for need to biopsy lesions classified with mammography, tomosynthesis (DBT) or ultrasound as 4A or 4B. CEM uses iodine contrast with dual low and high KeV mammogram images to create a contrast enhancement map of the breast that directly overlays the mammogram, thus providing anatomic and kinetic information, similar to MRI. The investigators found in a preliminary clinical trial that radiologists had higher true-positive rates and lower false-positive rates for biopsy recommendation with CEM than when using DBT and ultrasound. To validate those initial findings, the investigators propose to prospectively and sequentially perform CEM on 1855 consenting women with BIRADS 4A or 4B lesions detected on mammography, DBT or ultrasound. Prospectively radiologists will provide BIRADS ratings for every lesion using DBT alone, then with ultrasound and finally with CEM. With pathology known and based on the study design to minimize case by radiologist potential biases, the investigators plan to estimate the NPV level of CEM-based recommendations (overall and within the cases with conventionally confirmed biopsy recommendation) and demonstrate that it is sufficiently high, while leading to substantial reduction in biopsy recommendations for actually benign lesions. The investigators primary expectation is that the number of recommendations to biopsy benign lesions will decrease significantly (~20%), while maintaining high NPV (>95%) among the initial recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Subject is ≥30 years old
* Subject is diagnosed with a suspicious breast abnormality and is scheduled for an imaging directed breast biopsy.

Exclusion Criteria:

* Subject is unable or unwilling to undergo informed consent
* Subject has a breast implant in the breast of interest
* Subject is pregnant
* Subject is breast-feeding
* Subject is actively being treated for cancer of any type with chemotherapy
* Subject has reduced kidney function with eGFR < 30.
* Subject has had a prior reaction to iodinated contrast; thus a known allergy to iodinated contrast

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) | year 5
  The investigators will estimate and compare the changes in NPV of pre- and post CEM-based recommendations (where NPV is the proportion of pathology verified benign lesions out of post-CEM-downgraded to BIRADS 3 or lower).

SECONDARY OUTCOMES:
Positive Predictive Value of biopsies performed (PPV3) | year 5
  The investigators will estimate and compare the corresponding improvements in PPV3 in soft-tissue and calcification index-lesion cohorts.

OTHER OUTCOMES:
Frequencies | year 5
  The investigators will estimate the magnitude of the reduction in biopsies of benign soft-tissue index lesions (which approximates the increase in patient-level
Positive predictive value of biopsy recommendations (PPV2) | year 5
  The investigators will evaluate PPV of biopsy recommendations pre- and post-CEM by lesions' imaging appearance (mass, distortion, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Margarita L Zuley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Images may be shared with secondary investigators, including commercial companies after removal of all identifiers. All patient identification (name, patient number, birth date) will be removed from the DICOM headers of the images.
Time Frame: after publication for indefinitely
Access Criteria: secondary investigators for image analysis. Sharing via Box